CLINICAL TRIAL: NCT05185765
Title: An Application of Models Predicting the Eating Rate of Bread Using Sensory and Instrumental Texture
Acronym: BOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BOP.study
Record Dates: First submitted 2021-12-02; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Bread

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Brown bread (commercially available) (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread
- Wholemeal bread (commercially available) (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread
- Wholemeal bread without crust (commercially available) (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread
- White bread, water based (commercially available) (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread
- White hard roll (commercially available) (Active Comparator): Participants consume half a roll, and masticate and expectorate half of 1 cm thick slice
  Interventions: Other: Bread
- Brown hard roll (commercially available) (Active Comparator): Participants consume half a roll, and masticate and expectorate half of 1 cm thick slice
  Interventions: Other: Bread
- White soft bun (commercially available) (Active Comparator): Participants consume half a bun, and masticate and expectorate 1/8th of a bun
  Interventions: Other: Bread
- Brown soft bun (commercially available) (Active Comparator): Participants consume half a bun, and masticate and expectorate 1/8th of a bun
  Interventions: Other: Bread
- Ciabatta (commercially available) (Active Comparator): Participants consume half a mini ciabatta, and masticate and expectorate half of 1 cm thick slice
  Interventions: Other: Bread
- Croissant (commercially available) (Active Comparator): Participants consume half a croissant, and masticate and expectorate half of 1 cm thick slice
  Interventions: Other: Bread
- Whole wheat bread produced by bakery, proofing time 65 min, ambient cooling (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread
- Whole wheat bread produced by bakery, proofing time 85 min, ambient cooling (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread
- Whole wheat bread produced by bakery, proofing time 105 min, ambient cooling (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread
- Whole wheat bread produced by bakery, proofing time 65 min, vacuum cooling (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread
- Whole wheat bread produced by bakery, proofing time 85 min, vacuum cooling (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread
- Whole wheat bread produced by bakery, proofing time 105 min, vacuum cooling (Active Comparator): Participants consume half a slice, and masticate and expectorate 1/4th of rectangular bottom part
  Interventions: Other: Bread

INTERVENTIONS:
Other: Bread — Samples will be provided one by one labeled with an unique code. The mastication and expectorated sample will be given in replicate.

SUMMARY:
Rationale: The world-wide rising obesity rates are a major health problem. Therefore, people should moderate food intake. A lower eating rate will decrease the energy intake. The eating rate of foods can be modified by changing the texture without affecting their acceptability. Harder, chunkier, more viscous, and more voluminous foods will decrease the eating rate and thus energy intake. Bread is a staple food and contributes to a major part of the Dutch diet. By changing the proofing time and by applying vacuum cooling during the baking process, the texture of bread can be modified. The effect of this texture modification on eating rate is not investigated until now. To get an understanding of the relations between food texture and eating rate, modelling based on instrumental measurements is a promising technique as it can give valuable insights without sensorial and laboratorial labour and costs. However, it is not known if such a model can predict the eating rate as well as a model based on sensory measurements. Therefore, this study will investigate whether modelling of sensory or instrumental data predicts the eating rate of bread most accurate and can be applied for the product development of bread with modified eating rate.

Objective: The aim of the BOP-study is to compare mathematical models based on sensory or instrumental texture that predict the eating rate of bread and to validate if the models can be applied for the product development of bread with a modified eating rate by changing the proofing time and applying vacuum cooling.

Study design: The study consists out of a sensory study, instrumental measurements, and mathematical modelling. The sensory study is a randomised crossover trial. All participants consume all bread samples in a randomized order divided over four sessions. Every session will be video recorded.

Study population: Healthy Dutch adults (n=34) between 18-55 years old, and a BMI between 18.5-30 kg/m2 will be included.

Intervention: In the sensory study, participants will attend four test sessions during lunch in which sixteen bread samples will be investigated. Ten breads are commercially available and six breads are produced for product development purposes and differ in proofing time and vacuum cooling. In each session, a fixed portion of bread will be consumed by the participants during which the eating rate and sensory properties will be measured. Additionally, participants will chew and expectorate a bite-size piece of bread in replicate to determine the saliva addition to the bolus at time of swallowing.

Main study parameters/endpoints: The main study outcome is the eating rate (g/min).

ELIGIBILITY:
Inclusion Criteria:

* Good general health and appetite (self-report)
* Between 18-55 years old at the day of inclusion
* Dutch
* BMI 18.5-30 kg/m2 (self-report)
* Regular consumer of bread

Exclusion Criteria:

* Smoking
* Following a vegan diet
* Allergies or intolerance to any ingredient of the test meals
* Suffering from diabetes
* Having taste or smell disorders (self-report)
* Difficulties with swallowing, chewing and/or eating in general
* Use of medication that may influence study outcomes (self-report)
* Pregnant or lactating women
* Braces (not including a dental wire) or oral piercing
* Consuming on average more than 21 glasses of alcohol per week
* Not willing to stop using drugs during the study period (from inclusion till last test session)
* Men having facial hair such as a beard as facial movements cannot be analysed
* Signed up for participating in another research study
* Employee of Human Nutrition department of Wageningen University
* Employee, thesis student or intern at the chair group of Sensory Science and Eating Behaviour or Food Quality and Design (WUR)
* Don't like bread products

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Eating rate (g/min) | Up to 30 minutes
  Amount of the sample divided by the consumption time of the sample, measured with video recording

SECONDARY OUTCOMES:
Overall liking | Assessment will be done once every week for four weeks
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Crumb hardness | Assessment will be done once every week for four weeks
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Crumb dryness | Assessment will be done once every week for four weeks
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Crumb chewiness | Assessment will be done once every week for four weeks
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Crumb adhesiveness | Assessment will be done once every week for four weeks
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Crumb denseness | Assessment will be done once every week for four weeks
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Crust hardness | Assessment will be done once every week for four weeks
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Crust crispiness | Assessment will be done once every week for four weeks
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Crust crumbliness | Assessment will be done once every week for four weeks
  Measured using a 100-mm visual analogue scale (VAS) ranging from 'not at all' (0) to 'extremely' (100) with anchors at the beginning and end of the line
Bolus saliva content at moment of swallowing (g/g dry product) | Assessment will be done once every week for four weeks
  Participants will be instructed to chew on pieces of until they feel the urge to swallow. At this point the participants will expectorate the sample into an aluminium cup. Saliva content of the bolus at time of swallowing will be measured by dry matter content analysis. The boli are expectorated on aluminium dishes, weighted and dried for 24 h at 110 °C, and weighted again after drying. Bite-size pieces of each bread as given to the participants will be dried and weighted as well to determine the initial moisture content of the breads. The saliva content (g/g dry product) will be calculated by subtracting the initial moisture content of the bread from the moisture content of the bolus. The moisture content will be calculated based on a dry weight basis using MC= (m0 - m1)/m1, where m0 is the weight before drying and m1 is the weight after drying.

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No